CLINICAL TRIAL: NCT05326880
Title: Comparative Performance of Two-piece Zirconia Tissue Level Implants vs. Titanium Bone Level Implants Placed With a Fully Digital Workflow - 5-year Follow up of a Randomized Clinical Trial
Brief Title: 5-year Follow up Study on the Comparative Performance of Two-piece Zirconia and Titanium Implants
Acronym: PostNCT0390817
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Melissa Fok, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2022-03v1
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dental Implants; Single Tooth Lost; Dental Implant Failed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (SG) (Experimental): Receive new zirconia implant: Straumann® PURE 2-piece Ceramic Implant (tissue level), ZLA
  Interventions: Device: Ceramic Dental Implant
- Control Group (CG) (Active Comparator): Receive standard titanium implant: Straumann® Bone Level Implant, Titanium, SLA
  Interventions: Device: Titanium Dental Implant

INTERVENTIONS:
Device: Ceramic Dental Implant — The ceramic implant will be placed in healed extraction sockets in the premolar-to-premolar area in the mandible and maxilla for single tooth replacement followed by prosthetic loading with definitive prosthesis after 6 months healing time. Type 4 surgery will be performed as defined by the ITI Consensus Statements for Implant Placement in Extraction Sockets: healed sites, typically around 16 weeks after tooth was extracted or after tooth was lost to allow complete healing of the ridge as well as soft- and hard tissue maturation. Both SG and CG receive routine treatment, only the choice of the implant material is defined by the study protocol.
  Arms: Study Group (SG)
Device: Titanium Dental Implant — The titanium implant will be placed in healed extraction sockets in the premolar-to-premolar area in the mandible and maxilla for single tooth replacement followed by prosthetic loading with definitive prosthesis after 6 months healing time. Type 4 surgery will be performed as defined by the ITI Consensus Statements for Implant Placement in Extraction Sockets: healed sites, typically around 16 weeks after tooth was extracted or after tooth was lost to allow complete healing of the ridge as well as soft- and hard tissue maturation. Both SG and CG receive routine treatment, only the choice of the implant material is defined by the study protocol.
  Arms: Control Group (CG)

SUMMARY:
A post-market, randomized-controlled, superiority clinical study to compare medium-term performance and safety of the Straumann PURE 2-piece Ceramic Implant with Straumann Bone Level Implant using a fully digital workflow.

DETAILED DESCRIPTION:
Dental implants are a key modality for tooth replacement. Titanium dental implants have been the mainstay of dental implants as it osseointegrate well. Titanium has a silver gray metallic color and therefore, to hide its presence and enhance the aesthetic appearance, the implant is usually placed deeper into the bone tissue and the gums. This has negative consequences since it becomes more difficult to keep the interface between the dental implant and the crown free from bacterial plaque and inflammation. The use of zirconia（a base form of metal with similar properties of titanium in terms of osseointegration) has attracted a lot of interest because of its color that is similar to the one of natural teeth.This study will hence compare the long term performance of standard 4th generation dental implants made of titanium with a second generation zirconia dental implant. The study will evaluate the occurence of biological and technical complications; patient satisfaction and with the aesthetics of the tooth replacement over time.

ELIGIBILITY:
Inclusion Criteria:

following criteria must be met for inclusion in the study:

* Patients must have voluntarily signed the Informed Consent Form before any study related procedures are performed, are willing and able to attend scheduled follow-up visits and agree that the pseudonymized data will be collected, analyzed, and published.
* Patients must be males or females who are a minimum of 18 years of age.
* Patients, who have received a single tooth replacement with a study implant as per-protocol in the premolar-to-premolar area (excluding lower incisors) in the mandible and maxilla and restored with a screw retained ceramic crown.

Exclusion Criteria:

* Patients with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability.
* Pregnancy or intention to become pregnant at any point during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 60 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Bone level change | 5 years after implant loading (final crown restoration)
  Change in crestal bone level measured by analysis of standardized peri-apical xrays 5 years after loading [mm].

SECONDARY OUTCOMES:
Implant survival | 5 years after loading
  Implant survival rates 2, 3, 4, 5 years after loading: yes/no
Complication/event free survival | 5 years after loading
  To compare the complication/event free survival between two-piece ceramic implant and bone level titanium implant at 2, 3, 4, 5 years after loading.
14 item Oral Health Impact Profile (OHIP-14) | 5 years after loading
  The local language version of the OHIP-14 is a self-reported questionnaire that measures dysfunction, discomfort and disability attributed to oral conditions. The questionnaire focuses on seven dimensions of impact: Functional limitation; Pain; Psychological discomfort; Physical disability; Psychological disability; Social disability; Handicap. The patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4).

OTHER OUTCOMES:
Adverse Events | 5 years
  Adverse Events will be recorded at every visit throughout the observation period
Device Deficiencies | 5 years
  Any device complications and deficiencies will be recorded as Device Deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R. Fok, Dr., Principal Investigator — The University of Hong Kong
Locations (2):
- Dusseldorf University Hospital, Poliklinik für Zahnärztliche Prothetik, Düsseldorf, Germany
- Clinical Research Centre, Faculty of Dentistry, the University of Hong Kong, Hong Kong, Hong Kong